CLINICAL TRIAL: NCT02876848
Title: Adjuvant Endocrine Therapy in Breast Therapy in Breast Cancer: A Novel E-Health Approach in Optimizing Treatment for Seniors (OPTIMUM Study)
Brief Title: A Novel E-Health Approach in Optimizing Treatment for Seniors (OPTIMUM Study)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Ari Meguerditchian, Surgical Oncologist, McGill University Health Centre, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-37-2017-2535
Record Dates: First submitted 2016-08-16; First posted 2016-08-24 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Breast Neoplasms; Medication Adherence
Keywords: Administrative Claims, Healthcare; Aromatase Inhibitors; Breast Neoplasms; Health Services for the Aged; Medical Informatics Applications; Medication Adherence; Outcome and Process Assessment (Health Care); Selective Estrogen Receptor Modulators; Telemedicine
MeSH Terms: conditions — Breast Neoplasms; Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Site (Experimental): The hospital that will be the intervention site will have access to the OPTIMUM e-health tool. The intervention site cancer care team will receive the following OPTIMUM e-health alerts:
  1. An electronic alert of increased Adjuvant Endocrine Therapy discontinuation risk.
  2. An adherence to Adjuvant Endocrine Therapy monitor.
  3. An electronic discontinuation occurrence alert
  Interventions: Other: OPTIMUM e-health tool
- Control Site (No Intervention): The hospital that will be the control site will not have access to the OPTIMUM e-health tool. The cancer care team will continue to deliver care according to standard processes.

INTERVENTIONS:
Other: OPTIMUM e-health tool — If you are treated in a hospital that is using the OPTIMUM e-health tool ("intervention" group), once your care team receives any alerts, they may choose to:
  * Contact you over the phone or in person to provide medical advice on how to better take your pills,
  * Contact your pharmacist(s) and other doctors about your anti-cancer treatment.
  Arms: Intervention Site

SUMMARY:
Background: In women with hormone receptor positive (HR+) breast cancer, adjuvant endocrine therapy (AET) is associated with a significant survival advantage. Nonadherence is a particular challenge in older women, even though they stand to benefit the most from AET. Therefore, a novel e-health tool (OPTIMUM) that integrates real-time analysis of health administrative claims data was developed to provide point-of-care decision support for clinicians.

DETAILED DESCRIPTION:
Objectives: 1) To determine the effectiveness of a patient-specific, real-time e-health alerts delivered at point-of-care in reducing rates of AET discontinuation and to understand patient-level factors related to AET discontinuation. 2) To assess integration of e-health alerts regarding deviations from best practices in administration of AET by cancer care teams.

Methods: A prospective, two group controlled comparison pilot study will be conducted at two urban, McGill University-affiliated hospitals, the Royal Victoria Hospital and St. Mary's Hospital. A minimum of 43 patients per study arm will be enrolled through site-level allocation. Follow-up is 1.5 years. Healthcare professionals at the intervention site will have access to the e-health tool which will report to them in real-time: medical events with known associations to AET discontinuation, AET adherence monitor, and a discontinuation alert.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥ 65 years old,
2. Have been diagnosed with incident (non-metastatic) breast cancer,
3. Have a histologically-confirmed breast adenocarcinoma,
4. Have undergone breast surgery for stages I-III disease,
5. Have medical insurance with the Régie de l'Assurance Maladie du Québec (RAMQ) for at least 1 year prior to surgery,
6. Have HR positive disease,
7. Have no history of AET use prior to the diagnosis of breast cancer,
8. Expected to initiate AET or have only recently initiated AET (<6 months) but are free of previous discontinuation events,
9. Have the ability to consent for herself.

Exclusion Criteria:

male gender

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients discontinuing adjuvant endocrine therapy treatment | 1.5 years
  In each trial arm, the proportion of patients discontinuing AET treatment will be calculated as the number of patients discontinuing AET treatment divided by the total number of patients in that trial arm.

SECONDARY OUTCOMES:
Primary Non-adherence | 1.5 years
  In each trial arm, the proportion of patients who are prescribed AET treatment but do not fill any prescriptions will be calculated as the number of patients with primary non-adherence divided by the total number of patients in that trial arm.
Proportion of patients re-initiating after a discontinuation of adjuvant endocrine therapy treatment | 1.5 years
  In each trial arm, the proportion of patients re-initiating after a discontinuation of AET treatment will be calculated as the number of patients who start taking AET after a period of stopping divided by the total number of patients that discontinued in that trial arm.
Mean time to adjuvant endocrine therapy treatment re-initiation. | 1.5 years
  In each trial arm, mean time to AET treatment re-initiation will be calculated as the average number of days for a patient who has stopped taking AET treatment to start again, among those who start again (re-initiate).
Medical Possession Ratio ≥80% | 1.5 years
  In each trial arm, the proportion of patients that maintain a Medical Possession Ratio ≥80% will be calculated as the proportion patients whose proportion of number of days covered by medication supply in the treatment period is ≥80%.
Cancer Care Team Actions in the intervention arm - perform telephone follow-up with patient | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team called the patient will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the patient was called).
Cancer Care Team Actions in the intervention arm - perform telephone follow-up with community pharmacist | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team called the patient's pharmacist will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the patient's pharmacist was called).
Cancer Care Team Actions in the intervention arm - arrange for return to clinic with doctor | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team arranged for the patient to return to the clinic to see the doctor will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the cancer care team arranged a return to clinic with doctor).
Cancer Care Team Actions in the intervention arm - arrange for return to clinic with nurse | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team arranged for the patient to return to the clinic to see the nurse will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the cancer care team arranged a return to clinic with nurse).
Cancer Care Team Actions in the intervention arm - referral to doctor for closer follow-up | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team referred the patient to a doctor will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the cancer care team referred the patient to a doctor). Note that this action is different than the outcome "arrange for return to clinic with doctor" because this outcome occurs when a nurse directly schedules a patient to see a specific doctor without discussing with a doctor first.
Cancer Care Team Actions in the intervention arm - referral to cancer nurse for closer follow-up | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if a member of the cancer care team referred the patient to a cancer nurse will be assessed qualitatively (yes/no) and quantitatively (if yes, time in number of days before the cancer care team referred the patient to a cancer nurse).
Cancer Care Team Actions in the intervention arm - ignore the alert | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment, for that patient, if no action by the cancer care team was taken will be assessed qualitatively (yes/no) and quantitatively (how many alerts per patient were ignored). Note that "ignore the alert" is an explicit option that care teams can specify. They will be trained to understand that the "ignore the alert" option represents that the patient has not discontinued AET treatment and that they are of the opinion that the patient is not at risk of discontinuing AET treatment despite reading the alert.
Cancer Care Team Actions in the intervention arm - no changes in usual treatment despite new information provided | 1.5 years
  Upon alert receipt that a patient is at risk of discontinuing adjuvant endocrine therapy treatment or has discontinued AET treatment, for that patient, if no changes by the cancer care team were taken will be assessed qualitatively (yes/no) and quantitatively (how many alerts per patient were ignored). Note that this "no changes" is an explicit option that care teams can specify. They will be trained to understand that the "no changes" option represents that the patient requires other considerations beyond adhering to AET such as is stopping AET for upcoming surgery or no longer is indicated for AET based on disease progression (for e.g., brain metastases).
Cancer Care Team Actions in the intervention arm - Other | 1.5 years
  Any care team action that cannot be described by the predefined actions will be described by the care team in a free-text field for subsequent qualitative analysis. An overall theme or logical grouping of these qualitative outcomes will be explored and reported upon.

CONTACTS AND LOCATIONS:
Overall Officials: Ari N Meguerditchian, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Liane Feldman, MD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada